CLINICAL TRIAL: NCT01926535
Title: Comparative Analysis of Human Amniotic Membrane Graft Versus Contact Lenses in Syntomathic Bullous Keratopathy
Brief Title: Amniotic Membrane Graft In Syntomathic Bullous Keratopathy
Acronym: AMBUK
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Instituto para el Desarrollo Biotecnológico y la Innovación S.A. (Other); Universidad de Granada (Other)
Responsible Party: Principal Investigator, RICARDO ARIS, Interno de Medicina, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: RARIS-001
Record Dates: First submitted 2013-08-15; First posted 2013-08-21 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2013-08

CONDITIONS: Bullous Keratopathy
Keywords: amniotic membrane; contact lens; bullous keratopathy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Implant of amniotic membrane grafts (Experimental): Amniotic membrane grafts were implanted in the affected eyes using topical anesthesia. Each graft was sutured to the bulbar conjunctive tissue using 10-0 nylon sutures and a reinforcement stitch was applied at the cornea
  Interventions: Procedure: Implant of amniotic membrane grafts
- Therapeutic contact lenses (Active Comparator): Therapeutic contact lenses were applied in all patients and the lenses were replaced every two months according to the pre-established gold standard for this procedure.
  Interventions: Device: Therapeutic contact lenses

INTERVENTIONS:
Procedure: Implant of amniotic membrane grafts — Amniotic membrane grafts were implanted in the affected eyes using topical anesthesia. Each graft was sutured to the bulbar conjunctive tissue using 10-0 nylon sutures and a reinforcement stitch was applied at the cornea
  Arms: Implant of amniotic membrane grafts
Device: Therapeutic contact lenses — Therapeutic contact lenses were applied in all patients included in the control group and the lenses were replaced every two months according to the pre-established gold standard for this procedure.
  Arms: Therapeutic contact lenses

SUMMARY:
The amniotic membrane (AM) is an avascular structure derived from fetus, which is a good choice for regenerative medicine and effective treatment in eye surface pathologies such as bullous keratopathy (BK). This disease generates a chronic corneal edema evolving to the production of vesicles and bullae, chronic eye pain and visual acuity decrease.

Definitive treatment for those patients is corneal transplant; however, donation is not always available and thus requires long waiting times. The currently available palliative treatment consists in the use of contact lenses to prevent the corneal epithelium from falling. However, this may be associated with corneal neovascularization, lens displacement or loss, infections, and discomfort for the patient.

The objective of this work was to compare the use of amniotic membrane grafts versus contact lenses in patients suffering from BK awaiting a corneal transplant.

A randomized clinical trial assay was performed with patients with a clinical diagnosis of BK. Twenty patients were randomized into 2 groups: amniotic membrane and therapeutic contact lenses. Eye pain intensity (Analog visual scale), visual acuity (Snellen questioner), bullae and corneal epithelial defects presence, as well as corneal neovascularization and complications (biomicroscopy) were compared during 6 months.

DETAILED DESCRIPTION:
INTRODUCTION Handling of patients with severe eye surface injuries has always been challenging in the field of ophthalmology. One of the most significant pathologies causing severe injuries is Bullous Keratopathy (BK). This disorder is caused by a failure in corneal endothelial pump (Na+/K+/ATPase) characterized by chronic stromal edema, and it tends to evolve to the production of corneal vesicles and bullae due to the drainage of fluid to the anterior corneal layers as a consequence of intraocular pressure(1). Most common causes of BK are intraocular surgical procedures including those related to cataract surgery(2). This entity conforms the first cause for corneal transplant in the USA (from 26 to 50%) and the second in Europe(3,4,5).

Clinically, BK is characterized by chronic ocular pain, which is secondary to recurrent epithelial defects, ocular surface inflammation and visual sharpness decrease(1). Definitive treatment for patients with BK with remaining visual potential is corneal transplant. However, donor grafts are not always available and they often require long waiting times. For those reasons, medical and surgical palliative measures should be temporarily used to relief ocular pain. Among others, the use of therapeutic contact lenses stands out as one of the best alternatives due to its contribution to the prevention of epithelial falling and ulceration, acting as a mechanical bandage(6,7,8). These contact lenses do not improve visual sharpness neither contribute to the resolution of the problem that originated corneal edema. Besides, prolonged use of contact lenses may be associated to potential complications such as ocular disturbance, superficial neovascularization, inflammation and corneal infections, together with the economical expenses that patients have to deal with(6).

In 1940, De Roth described for the first time the use of human amniotic membrane (AM) in ophthalmology, and since that date, multiple studies guaranteed its application as an efficient treatment for ocular surface diseases(9,10, 11), including BK(12,13,14,15,16,17,18). AM is a thin membrane covering the foetal side of the placenta, and it consists of the external chorion (maternal origin) and the internal amnion (foetal origin). Histologically, it is composed of three layers: epithelium, basal membrane and stroma(19).

The therapeutic effect of the AM involves three basic synergistic actions on the ocular surface: 1) induction of growth and proliferation of new epithelia on the tissues (cornea and/or conjunctiva), 2) control of the inflammation of the tissues under the implant and 3) inhibition of fibrosis and neovascularization of the corneal stroma(19). For all these reasons AM might be an effective treatment to ameliorate disturbances generated by BK. In addition, human amniotic epithelial cells do not express HLA surface antigens, which justifies the absence of graft rejection in this type of transplants(20,21) and makes it a highly safe procedure.

In the present work, we describe the results of a randomized clinical trial in which the AM grafting technique was compared with the use of therapeutic contact lenses for the management of symptomatic bullous keratopathy in patients waiting for a corneal transplant at Carlos Van Buren Hospital from Valparaiso, Chile.

PATIENTS AND METHODS Study design Randomized clinical trial. Patients The universe of this clinical trial are all patients with clinical diagnosis of symptomatic bullous keratopathy (corneal bullae, recurrent eye pain, foreign body sensation and photophobia), diagnosed at the Department of Ophthalmology Hospital Carlos Van Buren, Valparaiso, Chile, who were on the waiting list for corneal transplant from January 2008 to October 2011. Excluded patients were those with medical contraindication to undergo surgery with topical anesthesia, patients with severe systemic conditions and patients with corneal infections.

Twenty patients, corresponding to universe of patients during this period, accepted to participate in this study and were included in this clinical trial. All patients provided written consent to participate in this study, and the trial was approved by the Ethics Committee of the Faculty of Medicine, Universidad de Valparaiso (Nº 10/2011). Patients were randomized on a simple random basis from a prefabricated list and divided into two groups: study group (N=10), with the implant of the AM, and control group (N=10), in which contact lenses were used.

Clinical data and variables considered for the study were: demography, etiology of BK, ocular pain (evaluated by using a visual analogue scale ranging from 0 to 10) and visual acuity (Snellen scale). By using a bio-microscope we evaluated the presence of bullae and epithelial defects per quadrant (with fluorescein test) and neovascularization. After treatment, the same equipment was used to check for presence of traces of AM and complications (infection, wound dehiscence, etc) through serial controls performed over a period of 6 months.

Interventions Human AM was prepared and preserved in the Biomedical Research Centre using a method previously described by Lee and Tseng (1995). In the study group, amniotic membrane (AM) grafts were implanted in the affected eyes using topical anesthesia. Each graft was sutured to the bulbar conjunctive tissue using 10-0 nylon sutures and a reinforcement stitch was applied at the cornea (Figure 1).

Therapeutic contact lenses were applied in all patients included in the control group and the lenses were replaced every two months according to the pre-established gold standard for this procedure.

Clinical follow-up examination was performed on days 1, 7, 30, and then monthly until 6 months for both groups. Both groups were managed with topical gentamicin each 4 hours during the first week after surgery.

Statistical analysis. Data were analysed with Stata SE 12.0 software. Results corresponding to continuous variables were described by medians and interquartile range (IQR) and categorical medians were described by percentages and frequencies. Mann-Whitney statistical test was used to detect statistical differences between two continuous variables, and Fisher exact test was used for categorical variables. Association between quantitative variables was established by Kendal's tau correlation test. For all analysis, a value of p<0.05 was considered statistically significant and all analyses were carried out double tailed.

ELIGIBILITY:
Inclusion Criteria:

All patients with clinical diagnosis of symptomatic bullous keratopathy (corneal bullae, recurrent eye pain, foreign body sensation and photophobia), diagnosed at the Department of Ophthalmology Hospital Carlos Van Buren, Valparaiso, Chile, who were on the waiting list for corneal transplant from January 2008 to October 2011

Exclusion Criteria:

Excluded patients were those with medical contraindication to undergo surgery with topical anesthesia, patients with severe systemic conditions and patients with corneal infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Ocular pain | 6 months
  Evaluated by using a visual analogue scale ranging from 0 to 10

SECONDARY OUTCOMES:
Visual acuity | 6 months
  Snellen scale
Corneal Neovascularization | 6 months
  Evaluation using a bio-microscope
Corneal epithelial defects | 6 months
  Evaluation using a bio-microscope per quadrant with fluorescein test
Complications | 6 months
  Evaluation using a bio-microscope

OTHER OUTCOMES:
Age | At the enrolling moment
  In years
Sex | At the enrolling moment
  Male or Female
Affected eye | At the enrolling moment
  left eye or right eye

CONTACTS AND LOCATIONS:
Overall Officials: L. Venegas, Principal Investigator — Ophthalmology Unit, Van Buren Hospital, Valparaiso, Chile.; M. Hettich, Principal Investigator — Ophthalmology Unit, Van Buren Hospital, Valparaiso, Chile.; J. Villena, Principal Investigator — Biomedical Research Centre, School of Medicine, Universidad de Valparaiso, Chile.; R. Aris, Principal Investigator — Biomedical Research Centre, School of Medicine, Universidad de Valparaiso, Chile.; M. Párraga, Principal Investigator — Biomedical Research Centre, School of Medicine, Universidad de Valparaiso, Chile.; O. Parolini, Principal Investigator — Centro di Ricerca E. Menni, Fondazione Poliambulanza-Istituto Ospedaliero, Brescia, Italy.; M. Alaminos, Principal Investigator — Department of Histology, University of Granada, Spain; A. Campos, Principal Investigator — Biomedical Research Centre, School of Medicine, Universidad de Valparaiso, Chile.; S, San Martin, Study Director — Biomedical Research Centre, School of Medicine, Universidad de Valparaiso, Chile.
Locations (1):
- Universidad de Valparaíso, Valparaíso, Región de Valparaíso, Chile

REFERENCES:
- [Background] Nishida T. Cornea: Fundamentals of cornea and external disease. St. Louis, Mosby. 1997; p. 3-27.
- [Background] Courtright P, Lewallen S, Holland SP, Wendt TM. Corneal decompensation after cataract surgery. An outbreak investigation in Asia. Ophthalmology. 1995 Oct;102(10):1461-5. doi: 10.1016/s0161-6420(95)30845-7. PMID 9097792
- [Background] Canner JK, Javitt JC, McBean AM. National outcomes of cataract extraction. III. Corneal edema and transplant following inpatient surgery. Arch Ophthalmol. 1992 Aug;110(8):1137-42. doi: 10.1001/archopht.1992.01080200117038. PMID 1497529
- [Background] Cosar CB, Sridhar MS, Cohen EJ, Held EL, Alvim Pde T, Rapuano CJ, Raber IM, Laibson PR. Indications for penetrating keratoplasty and associated procedures, 1996-2000. Cornea. 2002 Mar;21(2):148-51. doi: 10.1097/00003226-200203000-00003. PMID 11862083
- [Background] Maeno A, Naor J, Lee HM, Hunter WS, Rootman DS. Three decades of corneal transplantation: indications and patient characteristics. Cornea. 2000 Jan;19(1):7-11. doi: 10.1097/00003226-200001000-00002. PMID 10632000
- [Background] Jablonski J, Szafran B, Cichowska M. [Treatment of corneal complications after cataract surgery with soft contact lenses]. Klin Oczna. 1998;100(3):151-3. Polish. PMID 9813997
- [Background] Smiddy WE, Hamburg TR, Kracher GP, Gottsch JD, Stark WJ. Therapeutic contact lenses. Ophthalmology. 1990 Mar;97(3):291-5. doi: 10.1016/s0161-6420(90)32589-7. PMID 2336266
- [Background] Leibowitz HM, Rosenthal P. Hydrophilic contact lenses in corneal disease. II. Bullous keratopathy. Arch Ophthalmol. 1971 Mar;85(3):283-5. doi: 10.1001/archopht.1971.00990050285006. No abstract available. PMID 5542864
- [Background] Kim JC, Tseng SC. Transplantation of preserved human amniotic membrane for surface reconstruction in severely damaged rabbit corneas. Cornea. 1995 Sep;14(5):473-84. PMID 8536460
- [Background] Kim JC, Tseng SC. The effects on inhibition of corneal neovascularization after human amniotic membrane transplantation in severely damaged rabbit corneas. Korean J Ophthalmol. 1995 Jun;9(1):32-46. doi: 10.3341/kjo.1995.9.1.32. PMID 7674551
- [Background] Sangwan VS, Burman S, Tejwani S, Mahesh SP, Murthy R. Amniotic membrane transplantation: a review of current indications in the management of ophthalmic disorders. Indian J Ophthalmol. 2007 Jul-Aug;55(4):251-60. doi: 10.4103/0301-4738.33036. PMID 17595472
- [Background] Georgiadis NS, Ziakas NG, Boboridis KG, Terzidou C, Mikropoulos DG. Cryopreserved amniotic membrane transplantation for the management of symptomatic bullous keratopathy. Clin Exp Ophthalmol. 2008 Mar;36(2):130-5. doi: 10.1111/j.1442-9071.2008.01696.x. PMID 18352868
- [Background] Lee HI, Ha SW, Kim JC. A novel application of amniotic membrane in patients with bullous keratopathy. J Korean Med Sci. 2006 Apr;21(2):324-8. doi: 10.3346/jkms.2006.21.2.324. PMID 16614522
- [Background] Lopez Ferrando N, Celis Sanchez J, Gonzalez Del Valle F, Lopez Mondejar E. [Monolayered amniotic membrane transplantation as a palliative treatment for bullous keratopathy]. Arch Soc Esp Oftalmol. 2004 Jan;79(1):27-31. doi: 10.4321/s0365-66912004000100007. Spanish. PMID 14752699
- [Background] Espana EM, Grueterich M, Sandoval H, Solomon A, Alfonso E, Karp CL, Fantes F, Tseng SC. Amniotic membrane transplantation for bullous keratopathy in eyes with poor visual potential. J Cataract Refract Surg. 2003 Feb;29(2):279-84. doi: 10.1016/s0886-3350(02)01525-0. PMID 12648638
- [Background] Panda A, Pangtey MS, Sony P. Response to symptomatic management of postoperative bullous keratopathy with nonpreserved human amniotic membrane. Cornea. 2003 Mar;22(2):187; author reply 187-8. doi: 10.1097/00003226-200303000-00024. No abstract available. PMID 12605061
- [Background] Mejia LF, Santamaria JP, Acosta C. Symptomatic management of postoperative bullous keratopathy with nonpreserved human amniotic membrane. Cornea. 2002 May;21(4):342-5. doi: 10.1097/00003226-200205000-00002. PMID 11973379
- [Background] Pires RT, Tseng SC, Prabhasawat P, Puangsricharern V, Maskin SL, Kim JC, Tan DT. Amniotic membrane transplantation for symptomatic bullous keratopathy. Arch Ophthalmol. 1999 Oct;117(10):1291-7. doi: 10.1001/archopht.117.10.1291. PMID 10532436
- [Background] Shimmura S, Shimazaki J, Ohashi Y, Tsubota K. Antiinflammatory effects of amniotic membrane transplantation in ocular surface disorders. Cornea. 2001 May;20(4):408-13. doi: 10.1097/00003226-200105000-00015. PMID 11333331
- [Background] Adinolfi M, Akle CA, McColl I, Fensom AH, Tansley L, Connolly P, Hsi BL, Faulk WP, Travers P, Bodmer WF. Expression of HLA antigens, beta 2-microglobulin and enzymes by human amniotic epithelial cells. Nature. 1982 Jan 28;295(5847):325-7. doi: 10.1038/295325a0. No abstract available. PMID 6173762
- [Background] Akle CA, Adinolfi M, Welsh KI, Leibowitz S, McColl I. Immunogenicity of human amniotic epithelial cells after transplantation into volunteers. Lancet. 1981 Nov 7;2(8254):1003-5. doi: 10.1016/s0140-6736(81)91212-5. PMID 6118474
- See also: Link to the appropriate approved drug page at FDA's Drugs@FDA web site. — http://www.accessdata.fda.gov/scripts/cder/drugsatfda